CLINICAL TRIAL: NCT00205374
Title: Use of Cidofovir Injection in the Treatment of Recurrent Respiratory Papillomatosis."
Brief Title: Use of Cidofovir for Recurrent Respiratory Papillomatosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1999-196
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Recurrent Respiratory Papillomatosis
MeSH Terms: conditions — Recurrent respiratory papillomatosis | interventions — Cidofovir; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cidofovir (Active Comparator): Cidofovir (Vistide) is a commercially available agent approved by the FDA for the treatment of cytomegalovirus (CMV) retinitis in patients with acquired immunodeficiency syndrome (AIDS). The drug is not FDA approved for the treatment of RRP at this time. However, recent case reports have been encouraging with regard to the effectiveness of the agent in the treatment of RRP. The FDA has granted this study a "safe to proceed" designation with IND 58,481.
  Interventions: Drug: Cidofovir
- Placebo (Placebo Comparator): On the baseline study day, patients will be randomized into either a treatment group (cidofovir injection) or a placebo group. A restricted randomization procedure, in groups of 4, will be used to encourage uniformity in sample sizes between groups.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cidofovir — With regard to cidofovir concentration, the FDA has allowed us to inject a concentration of 5 mg/ml into both children and adults. The injection will add less than 2 additional minutes to the surgery time and discharge time will not be affected. Because the volumes of cidofovir injected into the airway will be reasonably small (typically less than 2 mL), the total systemic dose of cidofovir administered per visit will be far below the FDA-approved systemic limit of 5 mg/kg for HIV-related CMV retinitis.
  Other Names: Vistide
  Arms: Cidofovir
Drug: Placebo — On the baseline study day, patients will be randomized into either a treatment group (cidofovir injection) or a placebo group. A restricted randomization procedure, in groups of 4, will be used to encourage uniformity in sample sizes between groups.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
Recurrent respiratory papillomatosis (RRP) is the most common benign neoplasm of the larynx in the pediatric population. The impact of the disease on patients and families can be tremendous due to the need for frequent treatment. It would be highly beneficial to develop effective medical therapies as adjunctive measures to surgical ablation with the goal of reducing the frequency of reoccurrence.

DETAILED DESCRIPTION:
The focus of the present study is to evaluate the usefulness of cidofovir injection in diminishing the frequency and magnitude of papilloma recurrences in adult and pediatric RRP patients. Briefly, patients will be randomized into either a treatment (cidofovir injection) or a placebo group. The following measures will be made at each of 6 data collection time points, over the course of one year: (1) tumor load, based upon a published staging system for papilloma, (2) degree of respiratory obstruction for phonation, as assessed by phonation threshold pressures, and (3) general health, on validated health inventories (SF12 and Voice Handicap Index for adults; PedsQL (Trademarked) for children) and via measures of height weight and days absent from school or daycare, where applicable, for children. A repeated measures analysis will allow examination of time by treatment interactions to determine if the cidofovir injection group has fewer, or less severe, recurrences than the placebo group.

Specifically, we will answer the following questions in this investigation:

1. Does cidofovir injection reduce the frequency of RRP recurrences?
2. Does cidofovir injection reduce the magnitude of RRP, as assessed with a proposed staging system for RRP (Derkay et al., 1998) and measures of phonatory threshold pressure?
3. Does cidofovir injection improve general health, as assessed by height, weight and days absent from school in pediatric patients and health inventories (general health and voice-related) in children and adults?

ELIGIBILITY:
Inclusion Criteria:

* 4 surgeries for RRP in last 12 months

Exclusion Criteria:

* Renal insufficiency
* Nephrotoxic drugs in the last 7 days
* Sulfa allergies
* Currently treated with systemic or topical HPV chemotherapeutic agents
* Females of childbearing potential with a positive pregnancy test
* Women who are breast feeding

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 1999-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Scott McMurray, MD, Principal Investigator — University of Wisconsin Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McMurray JS, Connor N, Ford CN. Cidofovir efficacy in recurrent respiratory papillomatosis: a randomized, double-blind, placebo-controlled study. Ann Otol Rhinol Laryngol. 2008 Jul;117(7):477-83. doi: 10.1177/000348940811700702. PMID 18700421

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants in this randomized, double-blind, placebo-controlled clinical trial were 19 consecutive adult or pediatric patients who presented to the University of Wisconsin Otolaryngology-Head and Neck Surgery Clinic with a diagnosis of RRP who met inclusio/exclusion criteria and gave informed consent to participate.
Pre-assignment Details: Before inclusion in this study, and 48 hours before each cidofovir injection, laboratory tests confirmed that the (female) participants were not pregnant and that laboratory findings were not exclusionary for study participation.
Groups:
- Cidofovir: With regard to cidofovir concentration, the FDA has allowed us to inject a concentration of 5 mg/ml into both children and adults. The injection will add less than 2 additional minutes to the surgery time and discharge time will not be affected. Because the volumes of cidofovir injected into the airway will be reasonably small (typically less than 2 mL), the total systemic dose of cidofovir administered per visit will be far below the FDA-approved systemic limit of 5 mg/kg for HIV-related CMV retinitis. No more than 6 treatments were performed per patient within the 12-month time interval of the study.
- Placebo: The placebo treatment was injection of saline solution that had a color and viscosity identical to those of the active drug. Up to 6 injections per participant were given during the study.
Period: Overall Study
Arm/Group | Cidofovir | Placebo
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cidofovir; Placebo: On the baseline study day, patients will be randomized into either a treatment group (cidofovir injection) or a placebo group. A restricted randomization procedure, in groups of 4, will be used to encourage uniformity in sample sizes between groups.
- Total: Total of all reporting groups
Arm/Group | Cidofovir | Placebo | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (18) | 29 (12) | 31 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Papilloma Severity
Description: Derkay Severity Score. Minimum Score is Zero. Maximum score is 86. Treatment of RRP with cidofovir injection will be considered efficacious if drug group patients experience clinically or statistically significant changes in papilloma severity and inter-surgery time intervals (relative to pre-treatment assessments), when compared with placebo group patients.
  The scale rates - Voice (normal 0, abnormal 1, aphonic 2) Stridor (absent 0, present with activity 1, present at rest 2) Urgency of the intervention (scheduled 0, elective 1, urgent 2, emergent 3) Respiratory distress (none 0, mild 1, mod 2, severe 3, extreme 4).
  For multiple anatomical sites (18 or more) in the upper airway, left and right sides, lesions are rated as 0=none, 1=surface lesion, 2=raised lesion, and 3=bulky lesion).
  A higher rating value indicates more advanced disease and a worse outcome.
Time Frame: Baseline, 2 months, and 12 months
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Cidofovir | Placebo
Number analyzed (Participants) | 10 | 9
scores on a scale
  Baseline | 13.2 [5 to 33] | 12 [5 to 23]
  2 months | 3.7 [0 to 11] | 3.6 [1 to 11]
  12 months | 2.7 [0 to 13] | 5.1 [0 to 16]

2. Secondary Outcome: 12-month Change in Voice Handicap Index (VHI) Score
Description: Voice Handicap Index. This scale rates a patient's perception of voice related handicap in the domains of functional, physical, and emotional. There are 10 questions for each domain. Each question is rated by the subject on a 5-point scale, never =0, almost never =1, sometimes =2, almost always =3, always =4). A lower total score or domain score indicates improved, or less, voice handicap. Thus, the maximum total score is 4 X 30 = 120. For each domain, the maximum score is 4 X 10 = 40. Scores of 0 are the lowest possible score. In the paper we say that the Maximum score is 100, but obviously is it actually 120. Complete scale = 0-120.
  Lower score indicates improved perceived voice-realted quality of life.
Time Frame: 2 months, and 12 months
Population: [raw data no longer exist for this study, there a no data to report for a Baseline measure]
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | Cidofovir | Placebo
Number analyzed (Participants) | 10 | 9
scores on a scale
  2 months | 22 [0 to 59] | 32 [8 to 61]
  12 months | 31 [2 to 63] | 42 [0 to 93]

ADVERSE EVENTS:
Arm/Group | Cidofovir | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No